CLINICAL TRIAL: NCT03101410
Title: Gluten Sensibility in Elite Athletes
Acronym: GLUTHEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Institut Carnot Qualiment (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-308; 2016-A00356-45 (Other: 2016-A00356-45)
Record Dates: First submitted 2017-03-09; First posted 2017-04-05 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Intestinal Diseases; Gluten-sensitive
Keywords: Gluten; sport performance
MeSH Terms: conditions — Intestinal Diseases | interventions — Glutens; Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gluten (Experimental): Selected participants will be randomly allocated to treatment group (gluten or gluten free)
  Interventions: Behavioral: Gluten
- gluten fee (Experimental): Selected participants will be randomly allocated to treatment group (gluten or gluten free)
  Interventions: Behavioral: Gluten free

INTERVENTIONS:
Behavioral: Gluten — Selected participants will be randomly allocated to treatment group (gluten or gluten free).
  Arms: gluten
Behavioral: Gluten free — Selected participants will be randomly allocated to treatment group (gluten or gluten free).
  Arms: gluten fee

SUMMARY:
This clinical project aims to study the relationship between gluten consumption and its impact on digestive comfort, quality of life and performance of non-celiac athletes practicing an intensive physical activity..

DETAILED DESCRIPTION:
Gluten is a protein network that results from both, the hydration and the kneading of storage proteins contained in the endosperm of certain cereals. Gluten is particularly found in bread products but it is also found in many processed products because of its physicochemical properties (binding, swelling properties ...). This omnipresence is now blamed, and a growing percentage of the population reports "intolerance" to gluten. This gluten sensitivity hypothesis is frequently associated with intestinal disorders (irritable bowel syndrome, bloating, abdominal pain, chronic diarrhea, constipation) but also with headache, fatigue, muscle and joint aches, bone fragility, migraine, eczema, depression, anxiety .... This assumption has led to the adoption of increasingly frequent gluten-free diets among the general population, without medical justification.

Among the population, athletes are particularly concerned due to a higher prevalence of anaphylaxis dependent on the combination of physical exercise and food intake (Maulitz and Kidd syndrome). This syndrome is notably reported with consumption of cereals in particular wheat (bread, pasta). However, these conditions are poorly described with regards to gluten and scientific investigations are required to rationally characterize the benefits of gluten-free diets for elite athletes.

Therefore, this clinical project aims to study the relationship between gluten consumption and its impact on digestive comfort, quality of life and performance of non-celiac athletes practicing an intensive physical activity.

All the participants will give freely their written informed consent before their selection in the study.

Information on physical activities, demographics, anthropometrics, vital signs, relevant medical history and concomitant medication, dietary habits, usual dietary intake and nutritional supplements will be collected. All inclusion and exclusion criteria will be checked by the investigator or co-investigator.

Selected participants will be randomly allocated to treatment group (gluten or gluten free). Couple from the same family will be randomised in the same group.

After 2 months, all subjects will have the diet without gluten.

All recruited volunteers will be asked to replace their bread and pasta intake by study products (pasta and white bread with or without gluten), maintain their usual dietary habits and continue their normal physical habits.

Each 2 months, volunteers will have a physical performance assessment and will provide a blood and faeces samples. All volunteers will complete a follow-up questionnaire to obtain information about any changes in medication use, disease etc. Each week, all subjects will complete a questionnaire related to digestive function :Food Benefits Assessment (FBA)).

At the beginning and 2 months, usual dietary intakes will be estimated by means of a 3- days food records.

ELIGIBILITY:
Inclusion Criteria:

* Male and female trained >7h/week or more of 5 training/week
* Member of a sports federation or medical certificate fewer 3 months
* VO2 max estimated >125% of the theoretical value
* Regular consumption of gluten under different products
* Healthy (apparently free of diseases) and without any medical treatment
* Without digestive diseases and non-coeliac disease
* Affiliated to National Health Insurance
* Having normal capacity of training to enter in the study procedures
* Having provided her written informed consent

Exclusion Criteria:

* Medicals or surgical histories, evaluated non compatible by the investigator
* Diseases known
* Antibiotherapy 2 months before the study
* Gluten-free diet
* Individual unable to give informed consent or refusing to sign informed consent
* Being in exclusion on the National Volunteers Data file or refusing to be registered on the National Volunteers Data file
* Currently participating or who having got 4500€ in this year before to have participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Food Benefits Assessment (FBA) | at the beginning of the study, at 2 month and 4 month

SECONDARY OUTCOMES:
Physicals performances assessment : 3000m running performance | at the beginning of the study, at 2 month and 4 month
Microbiota composition analysis on faeces samples | at the beginning of the study, at 2 month and 4 month
  Microbiote composition will be measured by qPCR, targeting 16S gene
Changes in body composition measured by bioelectrical impedance | at the beginning of the study, at 2 month and 4 month
Qualities life index for digestive disorders modified (GIQLI assessment modified) | at the beginning of the study, at 2 month and 4 month
Inflammatory cytokines | at the beginning of the study, at 2 month and 4 month
Bone and joint cytokines | at the beginning of the study, at 2 month and 4 month
Immune function from lymphocytes | at the beginning of the study, at 2 month and 4 month
  Their reactivity will be studied in the presence of three different forms of gliadins: native, deaminated and hydrolysed

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France